CLINICAL TRIAL: NCT01508637
Title: Effect of Diesel Exhaust Exposures on Vascular Function in Humans: The Role of Sympathetic Activation
Brief Title: Diesel Exhaust and Vascular Function
Acronym: CVDTRAP4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joel Daniel Kaufman, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 39833-D; P50ES015915 (NIH)
Record Dates: First submitted 2012-01-05; First posted 2012-01-12 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Cardiovascular Effects
Keywords: air pollution; vasoconstriction; blood pressure; diesel exhaust
MeSH Terms: interventions — Vehicle Emissions; Terazosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diesel Exhaust + Terazosin (Experimental)
  Interventions: Other: Diesel Exhaust; Drug: Terazosin
- Diesel Exhaust + placebo (Experimental)
  Interventions: Other: Diesel Exhaust; Drug: placebo
- Filtered Air + terazosin (Sham Comparator)
  Interventions: Other: Filtered Air; Drug: Terazosin
- Filtered air + placebo (Sham Comparator)
  Interventions: Other: Filtered Air; Drug: placebo

INTERVENTIONS:
Other: Diesel Exhaust — Freshly generated diesel exhaust, diluted to 300 micrograms/cubic meter. Exposures are two hours in duration.
  Arms: Diesel Exhaust + Terazosin; Diesel Exhaust + placebo
Other: Filtered Air — Sham exposure, identical to conditions of diesel exhaust exposure, but with only air filtered of particles and volatile organic compound gases
  Arms: Filtered Air + terazosin; Filtered air + placebo
Drug: Terazosin — 2 mg by mouth, 90 minutes prior to exposure initiation
  Arms: Diesel Exhaust + Terazosin; Filtered Air + terazosin
Drug: placebo — capsule, identical in appearance to terazosin capsule, by mouth, 30 minutes prior to exposure initiation
  Arms: Diesel Exhaust + placebo; Filtered air + placebo

SUMMARY:
Double-blind, sham- and placebo-controlled randomized study of effects of freshly-generated diluted diesel exhaust inhalation on vascular function. To examine role of adrenergic system a trial of alpha-blocker terazosin is also used. Each participant completes four study sessions, separated by at least three weeks: 1) Diesel exhaust inhalation (DE, controlled at 300 micrograms/cubic meter for two hours) and terazosin (2 mg prior to inhalation exposure); 2) DE plus placebo (matched for terazosin); 3) filtered air plus terazosin; and 4) filter air plus placebo. The investigators assess outcomes of blood pressure, forearm brachial artery ultrasound, and plasma measures of endothelial activation. The investigators hypothesize that DE exposure will be associated with increased blood pressure, decreased brachial artery diameter, and increased circulating endothelins, and that these effects will be attenuated by terazosin administration.

ELIGIBILITY:
Inclusion Criteria:

* healthy without chronic illness
* Body Mass Index 18.5 - 26.0
* tolerates 2 mg terazosin dose without unacceptable symptoms
* able to return for four exposure sessions

Exclusion Criteria:

* any chronic disease
* tobacco user
* asthma
* elevated cholesterol
* obesity
* hypertension
* diabetes
* any chronic cardiovascular or pulmonary disease
* pregnancy or unwillingness to use effective contraception, if female

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 30-90 minutes after exposure initiation

SECONDARY OUTCOMES:
Brachial artery diameter | Assessed 30 minutes prior to exposure and 30 minutes post-exposure
  The investigators anticipate vasoconstriction (post-exposure vs. pre-exposure) as observed in this conduit artery in response to exposure to Diesel Exhaust, compared to Filtered Air sham exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Kaufman, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States